CLINICAL TRIAL: NCT02372448
Title: Multicenter Validation of the Sensitivity of Theranostic ALK Rearrangement Detection by FISH Analysis and Prevalence of Escaping Mutations in Circulating Tumor Cells for the Non-invasive Management of Lung Cancer Patients
Acronym: STALKLUNG01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-APN-01
Record Dates: First submitted 2014-09-22; First posted 2015-02-26 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALK-positive (Other): ALK positive analysis on CTCs detected by ISET
  Interventions: Other: ALK analysis on CTCs detected by ISET
- ALK-negative (Other): ALK negative analysis on CTCs detected by ISET
  Interventions: Other: ALK analysis on CTCs detected by ISET

INTERVENTIONS:
Other: ALK analysis on CTCs detected by ISET

SUMMARY:
Patients eligibility to targeted therapies relies on a molecular test performed on a tumor sample collected by biopsy. This invasive procedure is associated with a relative high risk of morbidity and requires the intervention of a costly and important technical platform. Thus, inoperable patients can be deprived from potentially more efficient therapies. A "liquid biopsy" of Circulating Tumor Cells (CTCs) present in the blood and their molecular characterization is an appealing alternative to meet an urgent need for these patients. Moreover no CTC-based molecular test is currently routinely available.

The 5-year survival rate of patients with non-small cell lung carcinoma (NSCLC) is low. Recent reports demonstrated that the detection of an ALK rearrangement in the tumor tissue allows patients with late-stages NSCLC to benefit from crizotinib treatment.

However, 1) the detection of an ALK rearrangement is currently performed on small biopsies or fine-needle aspirates and can be hindered by the limited tissue quantities available. Tumor tissue is difficult to obtain in patients with advanced/metastatic lung cancer for whom surgery is rarely a component of treatment. Finding alternative and more effective means of diagnosing an ALK rearrangement are critical issues for identifying patients who may benefit from treatment with crizotinib; 2) some patients develop resistance to crizotinib due to de novo ALK mutations.

In this setting, circulating tumor cells (CTCs), which have been shown to be detectable by ISET (Isolation by Size of Epithelial Tumor Cells) method in 80% to 100 % of late stages lung cancer patients represent a non-invasive and easily accessible source of tumor material for assessing ALK rearrangement and escaping mutations in a kinetic manner. The ISET method was first published in 2000 and several independent teams have now established its high sensitivity and specificity of ISET for NSCLC. With ISET, specificity can be achieved using the same methods and criteria used by cytopathologists to diagnose solid tumors.

The high sensitivity and specificity of ISET are two essential starting points for the feasibility of this present project. Low-throughput molecular characterization of CTCs isolated by ISET has also been achieved. The remaining challenge consists in developing high-throughput ISET-based molecular tests for personalized medicine that are transferable to the clinics.

The Team 1 at the CHU de Nice and the Team 2 at the Gustave Roussy Institute have demonstrated that the detection of an ALK rearrangement in CTC isolated by ISET is feasible and consistent with results obtained in corresponding tumor tissues. In this context, the aim of this project is to obtain 1) a definitive prospective clinical validation of the use of CTC as an alternative to tumor tissue for ALK analysis-based patients stratification; 2) a proof that escaping mutations can be detected early by kinetic analysis of CTC in patients treated by crizotinib. ALK rearrangement will be prospectively investigated in CTCs isolated by ISET at diagnosis and during follow up from patients with stage IIIb/IV lung cancer and de novo mutations will be searched in patients with resistance to crizotinib. This study will provide both clinical and economic benefit to targeted treatment of patients with advanced lung cancer.

This project is strongly original as no CTC-based ALK rearrangement test has been independently validated up to now with clinical samples. The development of non-invasive theranostic test through the genetic analysis of CTCs is a clinically relevant goal for non-invasive stratification of cancer patients, avoiding morbidity related to lung biopsy and surgery. It would allow determining patient's eligibility to targeted therapies on a blood sample analysis. CTC-based ALK test could be useful to guide the choice of ALK targeted therapy in patients with lung cancer. Furthermore, developing biomarkers based on CTCs analysis would open the way to the non-invasive follow up of aggressive cancers, early detection of mutations associated with resistance to targeted therapies and tailoring treatment to a real time analysis of the evolving tumor cell populations. This test is expected to markedly improve patients' quality of life avoiding invasive diagnostic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Histologically confirmed stage IIIb/IV non-squamous NSCLC undergoing biopsy or surgery
* Presence of ALK rearrangement result by FISH analysis (gold standard method) on tumor tissue
* Signed specific informed consent approved by the Institutional Review Board prior to patient entry
* Affiliation to the social security system

Exclusion Criteria:

* Vulnerable persons: adults under guardianship or persons deprived of their liberty, patients under 18 years old
* Medical and/or psychiatric problems of sufficient severity to limit full compliance with the study or expose patients to undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
sensitivity and specificity of the FISH technique for the detection of the ALK rearrangement in CTCs Change from Baseline to 6 and 12 months | at the inclusion, 6 months and 12 months
  ALK rearrangement positivity by FISH analysis in CTC will be defined as the presence of an ALK rearrangement in four or more CTCs isolated per 1 ml blood. The proportion of ALK-rearranged CTCs (determined by FISH analysis) among the total numbers of CTCs determined by cytomorphological examination or by combining immunofluorescent staining and cytomorphological examination will be also determined and compared to that obtained in the tumor tissue.

SECONDARY OUTCOMES:
sensitivity and specificity of the ICC analysis on CTCs | at the inclusion, 6 months and 12 months
  The intensity of cytoplasmic staining as well as percentages of positive CTCs will be assessed as follows: 0 = no or faint staining in <10% CTCs; 1+ = faint staining in >10% CTCs; 2+ = moderate staining in >10% CTCs; 3+ = strong staining in >10% CTCs. Positive ALK expression is considered as between 2+ and 3+.
association between the ALK-rearranged CTC levels evolution and tumor progression at 6 and 12 months | at the inclusion, 6 and 12 months
  The ALK-rearranged CTC levels evolution will be defined as the difference, between baseline and respectively M6 and M12, of the CTC number per 1 ml blood as determined by the ISET method. The systemic progression under crizotinib or another ALK inibitor will be evaluated according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 (http://www.recist.com/). Patients will be categorized into 3 groups with: stable disease, response (complete/partial) or with progressive disease. The association will be adjusted on covariates such as gender, age, smoking history, histology, T4 subtypes (in patients with stage IIIB), and M1 subtypes (in patients with stage IV disease), the initial treatment modality (i.e., surgery, radiotherapy, none, or both).

CONTACTS AND LOCATIONS:
Overall Officials: Paul HOFMAN, Pr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (11):
- France (11):
  - Centre François Baclesse, Caen
  - Grenoble university hospital, Grenoble
  - Marseille University Hospital, Marseille
  - Nancy university hospital, Nancy
  - Centre Antoine Lacassagne, Nice
  - CHU de Nice, Nice
  - Hôpital Tenon, Paris
  - Institut arnault tzanck, Saint-Laurent-du-Var
  - Toulouse University Hospital, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif